CLINICAL TRIAL: NCT04235621
Title: A Study to Characterize the Genetic, Biomarker, and Clinical Profile of Patients With Focal Segmental Glomerulosclerosis (FSGS), Treatment-Resistant Minimal Change Disease (TR-MCD), and Diabetic Nephropathy (DN)
Brief Title: A Study to Understand the Genetics and Clinical Course of Focal Segmental Glomerulosclerosis (FSGS), Treatment-Resistant Minimal Change Disease (TR-MCD), and Diabetic Nephropathy (DN)
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision for administrative reasons
Sponsor: Goldfinch Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GFB-887-501
Record Dates: First submitted 2019-12-31; First posted 2020-01-22 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Glomerulosclerosis, Focal Segmental; Minimal Change Disease; Diabetic Nephropathies
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FSGS/TR-MCD: Patients with FSGS/TR-MCD
  Interventions: Other: FSGS/TR-MCD
- Diabetic Nephropathy (DN): Patients with DN
  Interventions: Other: Diabetic Nephropathy (DN)

INTERVENTIONS:
Other: FSGS/TR-MCD — This is a non-interventional study
  Groups: FSGS/TR-MCD
Other: Diabetic Nephropathy (DN) — This is a non-interventional study
  Groups: Diabetic Nephropathy (DN)

SUMMARY:
This is a study with 2 parts. Part 1 comprises a visit to collect biological samples necessary for the molecular characterization of chronic kidney disease. Part 2 comprises an observational period of 5 visits over a period up to 8 weeks. During Part 2, baseline tests will be conducted, and urine will be collected approximately every 2 weeks for 8 weeks. Patients may participate in Part 1, Part 2, or both, and will be followed for up to 1 year consisting of data collection from the patient's medical records and home collection of urine samples every 4 months.

ELIGIBILITY:
Inclusion Criteria:

For FSGS/TR-MCD patients :

1. Competent and willing to provide informed consent and adhere to all study assessments and restrictions.
2. Male or female ≥ 18 years of age with FSGS or TR-MCD at the time of providing written informed consent.
3. Diagnosis of FSGS or TR-MCD, based on either biopsy or genetic testing.
4. Urinary protein to creatinine ratio (UPCR) ≥ 1.0 g/g.
5. Estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2.

For DN patients:

1. Competent and willing to provide informed consent and adhere to all study assessments and restrictions.
2. Male or female ≥ 18 years of age with DN at the time of providing written informed consent.
3. Diagnosis of type 2 diabetes
4. Urinary albumin to creatinine ratio (UACR) ≥ 150 mg/g.
5. Estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2.

Exclusion Criteria:

For FSGS/TR-MCD patients:

1. Evidence of another kidney disease or kidney disease secondary to an infectious process.
2. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. Patients whose results are compatible with prior immunization or treatment may be included.
3. Body mass index (BMI) > 42 kg/m2.
4. Significant history or evidence of clinically significant disorder, condition, current illness, or disease that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion (eg, severe cardiac disease, cardiac conduction defect, or severe or chronic hepatobiliary disease).
5. History of malignancy not in remission within the last 5 years other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
6. History of any organ or bone marrow transplant, including kidney grafts.
7. History of alcoholism or drug/chemical abuse within 12 months.
8. Preplanned surgery or procedures that would interfere with the conduct of the study.

For DN patients:

1. Evidence of another kidney disease or kidney disease secondary to an infectious process.
2. History of HIV, hepatitis B, or hepatitis C. Patients whose results are compatible with prior immunization or treatment may be included.
3. BMI > 42 kg/m2.
4. Significant history or evidence of clinically significant disorder, condition, current illness, or disease that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion (eg, severe cardiac disease, cardiac conduction defect, or severe or chronic hepatobiliary disease).
5. History of malignancy not in remission within the last 5 years other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
6. History of any organ or bone marrow transplant, including kidney grafts.
7. History of alcoholism or drug/chemical abuse within 12 months.
8. Preplanned surgery or procedures that would interfere with the conduct of the study.
9. Renal disease that requires immunosuppressive therapy (currently, or in the past).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be drawn from participating investigators' clinics
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Change in Urine Protein-to-Creatinine Ratio (UPCR) | Approximately 1 year
Change in Urine Albumin-to-Creatinine Ratio (UACR) | Approximately 1 year
Estimated Glomerular Filtration Rate (eGFR) | Baseline/Biomarker collection visit
Change in Estimated Glomerular Filtration Rate (eGFR) | Approximately 8 weeks
Change in Urine Biomarker: Nephrin | Approximately 1 year
Change in Urine Biomarker: Podocin | Approximately 1 year
Change in Urine Biomarker: Rac1 | Approximately 1 year
Change in Urine Biomarker: Synaptopodin | Approximately 1 year
Change in Urine Biomarker: Urea | Approximately 1 year
Change in Urine Biomarker: Other Exploratory | Approximately 1 year
Change in Serum/Plasma Biomarker: Other Exploratory | Approximately 8 weeks
Number of patients with genetic variants predicted to be associated with chronic kidney disease and functional consequence | Baseline/Biomarker collection visit
  DNA analysis of blood sample
Gene expression profile and phenotype of inducible pluripotent stem cell (iPSC)-generated organoids | Baseline/Biomarker collection visit
  Generation of iPSC from whole blood sample
Change from Baseline Patient-reported Assessment of FSGS Symptoms | Approximately 8 weeks
  FSGS/TR-MCD patients will assess disease symptomatology utilizing the FSGS Symptom Diary and FSGS Symptom Impact Questionnaire
Change from Baseline Patient-reported Assessment of Health Status | Approximately 8 weeks
  Patients will assess health status using the 36-Item Short Form Health Survey (SF-36)
Change from Baseline Patient-reported Assessment of Fatigue | Approximately 8 weeks
  Patients will assess the symptom of fatigue utilizing the Modified Fatigue Impact Scale
Change from Baseline Clinician-reported Assessment of Edema | Approximately 8 weeks
  Clinicians will assess edema in FSGS/TR-MCD patients using a standardized measurement of edema in FSGS/TR-MCD patients
Incidence of Untoward Medical Occurrences | Approximately 1 year
  Incidence of untoward medical occurrences that result in death; are life threatening; require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; or result in an important medical event.
% of Patients with Change in Treatment | Approximately 1 year
  Change in treatment as indicated by patient medical record

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Aventiv Research - Phoenix, Mesa, Arizona
  - Glendale Adventist Medical Center, Glendale, California
  - DaVita Mojave Sage Dialysis, Victorville, California
  - Colorado Kidney Care, Denver, Colorado
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - St. Clair Nephrology, Roseville, Michigan
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Clinical Research Consultants, Kansas City, Missouri
  - DaVita Pelican Point Dialysis, Las Vegas, Nevada
  - High Desert Nephrology, Gallup, New Mexico
  - Akron Nephrology Associates, Inc., Akron, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Arlington Nephrology, PC, Arlington, Texas
  - North Texas Kidney Disease Association, Lewisville, Texas
  - South Texas Renal Care Group (Downtown), San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group (Wurzbach Road), San Antonio, Texas
  - South Texas Renal Care Group (Westover Hills), San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group (Carnoustie Drive), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient reported outcome (and other relevant data) will be shared with other researchers.